CLINICAL TRIAL: NCT00878618
Title: A Phase I, Single-Centre, Open, Randomized, Two-Way Crossover Study to Evaluate the Pharmacokinetics of the Extended-Release Test Formulation of AZD0837 Compared to the Extended-Release AZD0837 Reference Formulation After Repeated Dosing in Healthy Volunteers
Brief Title: Pharmacokinetics of Extended-Release Test- and Reference Formulations of AZD0837
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Karin Wåhlander, Medical Science Director, AstraZeneca R&D Mölndal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1250C00056
Record Dates: First submitted 2009-03-31; First posted 2009-04-09 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — AZD 0837

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HAB (Experimental): AZD0837 test- (in session 1) and reference- (in session 2) formulation with heavy breakfast
  Interventions: Drug: AZD0837
- HBA (Experimental): AZD0837 reference- (in session 1) and test- (in session 2) formulation with heavy breakfast
  Interventions: Drug: AZD0837
- LAB (Experimental): AZD0837 test- (in session 1) and reference- (in session 2) formulation with light breakfast
  Interventions: Drug: AZD0837
- LBA (Experimental): AZD0837 reference- (in session 1) and test- (in session 2) formulation with light breakfast
  Interventions: Drug: AZD0837

INTERVENTIONS:
Drug: AZD0837 — Extended-release tablets, test formulation. 2 tablets given in the morning for 6 days
  Arms: HAB; LAB
Drug: AZD0837 — Extended-release tablets, reference formulation. 2 tablets given in the morning for 6 days
  Arms: HBA; LBA

SUMMARY:
The aims of this study are to evaluate the pharmacokinetics, safety and tolerability of the oral doses of the extended-release test- and reference formulations of AZD0837 in healthy volunteers both in fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject aged between 18 to 45 years inclusive
* Body mass index (BMI) between 19 to 30 kg/m2 inclusive
* Body weight between 50 to 100 kg inclusive
* Women must be either post-menopausal, permanently sterilised or, if of childbearing potential, must have a negative pregnancy test before intake of study medication and use a reliable form of contraception before and during participation in the study.

Exclusion Criteria:

* Significant illness (including ongoing or history of liver disease), trauma or surgical procedures from 2 weeks before the pre-entry visit until the first administration of Investigational Product
* Clinical significant abnormalities in clinical chemistry, haematology or urinalysis result including positive result on screening tests for serum hepatitis B surface antigen, hepatitis C antibody or HIV or positive F-Hb result pre-entry
* History of bleeding disturbance (including extensive menstrual bleedings) or thrombotic disorder
* Clinically significant medical history, as judged by the investigator, including psychiatric disorders or severe allergies.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-04; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of AZD0837 and the active metabolite AR-H067637XX for the extended-release test formulation of AZD0837 compared to the ER reference formulation. | Intense PK-sampling during 5 pre- defined study days for PK profiling. In 2 of the study days the subjects will have a breakfast before intake of the Investigational Product.

SECONDARY OUTCOMES:
To evaluate the PK of the intermediate metabolite AR-H069927XX | Since the metbolite will be evaluated from the AZD0837-samples the time frame is the same as above.
Safety variables (ECG, pulse, blood pressure, safety lab, physical examination, adverse events) | ECG & physical examination at start and end of study. Pulse and blood pressure predose day 1 and every day 2 h post dose. Adverse events collected during the whole study. Safety lab at a few timepoints but APTT will be checked on 4 h post dose on day 1.
Measurement of plasma concentrations of 4 beta-hydroxycholesterol to investigate whether AZD0837 affects the level of CYP3A4 | Once predose on day 1, session 1 and once predose on day 5, session 2

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Edén Eden, Principal Investigator — Quintiles AB, Uppsala, Sweden
Locations (1):
- Research Site, Uppsala, Sweden